CLINICAL TRIAL: NCT04650854
Title: An Open-Label Extension Study to Evaluate Rozanolixizumab in Study Participants With Generalized Myasthenia Gravis
Brief Title: A Study to Evaluate Rozanolixizumab in Study Participants With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0007; 2020-003230-20 (EudraCT Number)
Record Dates: First submitted 2020-11-05; First posted 2020-12-03 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Generalized Myasthenia Gravis
Keywords: UCB7665; generalized myasthenia gravis; rozanolixizumab; gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rozanolixizumab dosage regimen 1 (Experimental): Study participants randomized/assigned to dosage regimen 1 will receive assigned dosage of rozanolixizumab for the initial cycle. The dose regimen may be switched before the start of each subsequent treatment cycle based on investigator discretion.
  Interventions: Drug: Rozanolixizumab
- Rozanolixizumab dosage regimen 2 (Experimental): Study participants randomized/assigned to dosage regimen 2 will receive assigned dosage of rozanolixizumab for the initial cycle. The dose regimen may be switched before the start of each subsequent treatment cycle based on investigator discretion.
  Interventions: Drug: Rozanolixizumab

INTERVENTIONS:
Drug: Rozanolixizumab — Rozanolixizumab will be administered by subcutaneous infusion in dosage regimen 1 or 2.
  Other Names: UCB7665

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of additional 6-week treatment cycles with rozanolixizumab in study participants with generalized myasthenia gravis (gMG).

ELIGIBILITY:
Inclusion Criteria:

* Study participant must meet one of the following:

  1. completed MG0003 [NCT03971422]
  2. required rescue therapy during the Observation Period in MG0003 or
  3. completed at least 6 visits in MG0004 [NCT04124965]
* Body weight ≥35 kg at Baseline (Day 1)
* Study participants may be male or female

Exclusion Criteria:

* Study participant has a known hypersensitivity to any components of the study medication or other anti-neonatal Fc receptor (FcRn) medications
* Study participant with a known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent tuberculosis infection (LTBI), or current/history of nontuberculous mycobacterial infection (NTMBI)
* Study participant met any mandatory withdrawal or mandatory study drug discontinuation criteria in MG0003, or MG0004, or permanently discontinued study drug in either study
* Study participant intends to have a live vaccination during the course of the study or within 8 weeks following the final dose of rozanolixizumab
* Study participant with severe (defined as Grade 3 on the Myasthenia Gravis-Activities of Daily Living (MG-ADL) scale) weakness affecting oropharyngeal or respiratory muscles, or who has myasthenic crisis or impending crisis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 22733 (UCB)
Locations (69):
- United States (13):
  - Mg0007 50092, Orange, California
  - Mg0007 50099, San Francisco, California
  - Mg0007 50122, Miami, Florida
  - Mg0007 50120, Miami, Florida
  - Mg0007 50073, Tampa, Florida
  - Mg0007 50075, Augusta, Georgia
  - Mg0007 50323, Honolulu, Hawaii
  - Mg0007 50114, Indianapolis, Indiana
  - Mg0007 50121, Lexington, Kentucky
  - Mg0007 50077, New York, New York
  - Mg0007 50090, Winston-Salem, North Carolina
  - Mg0007 50096, Philadelphia, Pennsylvania
  - Mg0007 50113, Houston, Texas
- Canada (5):
  - Mg0007 50071, Edmonton
  - Mg0007 50066, Montreal
  - Mg0007 50124, Montreal
  - Mg0007 50070, Québec
  - Mg0007 50069, Toronto
- Czechia (2):
  - Mg0007 40125, Ostrava - Poruba
  - Mg0007 40124, Prague
- Denmark (3):
  - Mg0007 40128, Aalborg
  - Mg0007 40127, Aarhus
  - Mg0007 40126, Copenhagen
- France (5):
  - Mg0007 40129, Bordeaux
  - Mg0007 40360, Limoges
  - Mg0007 40132, Nice
  - Mg0007 40133, Paris
  - Mg0007 40131, Strasbourg
- Georgia (5):
  - Mg0007 20160, Tbilisi
  - Mg0007 20161, Tbilisi
  - Mg0007 20163, Tbilisi
  - Mg0007 20164, Tbilisi
  - Mg0007 20165, Tbilisi
- Germany (5):
  - Mg0007 40134, Essen
  - Mg0007 40140, Göttingen
  - Mg0007 40139, Jena
  - Mg0007 40078, Leipzig
  - Mg0007 40177, Münster
- Italy (6):
  - Mg0007 40283, Bologna
  - Mg0007 40144, Milan
  - Mg0007 40307, Napoli
  - Mg0007 40146, Pavia
  - Mg0007 40148, Roma
  - Mg0007 40150, Roma
- Japan (10):
  - Mg0007 20035, Bunkyō City
  - Mg0007 20068, Chiba
  - Mg0007 20078, Hanamaki-shi
  - Mg0007 20079, Hiroshima
  - Mg0007 20075, Kobe
  - Mg0007 20071, Nagasaki
  - Mg0007 20077, Sendai
  - Mg0007 20070, Shinjuku-ku
  - Mg0007 20076, Shinjuku-ku
  - Mg0007 20032, Suita
- Poland (4):
  - Mg0007 40155, Gdansk
  - Mg0007 40154, Lodz
  - Mg0007 40151, Lublin
  - Mg0007 40153, Poznan
- Russia (4):
  - Mg0007 20169, Novosibirsk
  - Mg0007 20001, Saint Petersburg
  - Mg0007 20028, Saint Petersburg
  - Mg0007 20055, Saint Petersburg
- Mg0007 40467, Niš, Serbia
- Spain (4):
  - Mg0007 40160, Barcelona
  - Mg0007 40157, L'Hospitalet de Llobregat
  - Mg0007 40350, Murcia
  - Mg0007 40308, San Sebastián de los Reyes
- Taiwan (2):
  - Mg0007 20081, Taipei
  - Mg0007 20086, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Derived] Bril V, Druzdz A, Grosskreutz J, Habib AA, Kaminski HJ, Mantegazza R, Sacconi S, Utsugisawa K, Vu T, Boehnlein M, Gayfieva M, Greve B, Woltering F, Vissing J; MG0004 study investigators. Safety and efficacy of chronic weekly rozanolixizumab in generalized myasthenia gravis: the randomized open-label extension MG0004 study. J Neurol. 2025 Mar 19;272(4):275. doi: 10.1007/s00415-025-12958-9. PMID 40105996
- [Derived] Bril V, Druzdz A, Grosskreutz J, Habib AA, Mantegazza R, Sacconi S, Utsugisawa K, Vissing J, Vu T, Boehnlein M, Bozorg A, Gayfieva M, Greve B, Woltering F, Kaminski HJ; MG0003 study team. Safety and efficacy of rozanolixizumab in patients with generalised myasthenia gravis (MycarinG): a randomised, double-blind, placebo-controlled, adaptive phase 3 study. Lancet Neurol. 2023 May;22(5):383-394. doi: 10.1016/S1474-4422(23)00077-7. PMID 37059507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in February 2021 and concluded in January 2024. Participant Flow refers to Full Analysis Set (FAS).
Pre-assignment Details: Participants who completed MG0003 (NCT03971422) or required rescue therapy during Observation Period (OP) in MG0003 (except for participants who received intravenous immunoglobulin/plasma exchange in MG0003) or completed at least 6 treatment visits in MG0004 (NCT04124965) were enrolled in this study.
Groups:
- Enrolled, But Not Treated: Participants were enrolled but did not receive a treatment cycle of Rozanolixizumab (RLZ) in MG0007 per the Investigator's discretion.
- Rozanolixizumab ~7 mg/kg: Eligible participants from MG0003 were randomized to receive an initial fixed 6-week treatment cycle of subcutaneous (sc) dose of Rozanolixizumab (RLZ) equivalent to approximately 7 milligrams/kilogram (mg/kg) once weekly (QW), followed by OP that began after last dose of that treatment cycle. Eligible participants from MG0004 who completed at least 6 scheduled visits for RLZ treatment, premature end of treatment (PEOT) Visit and who were in OP could complete End of Study Visit could move directly into OP in MG0007. These participants underwent their first MG0007 treatment with RLZ upon worsening of MG symptoms. Participants continued their last treatment dose from MG0004. Dose adjustments could be applied in further cycles as per Investigator's discretion. If symptom worsens between assessments, resulting in need for additional treatment, participants underwent another 6-week treatment cycle followed by OP, based on Investigator's discretion.
- Rozanolixizumab ~10 mg/kg: Eligible participants from MG0003 were randomized to receive an initial fixed 6-week treatment cycle of sc dose of RLZ equivalent to approximately 10 mg/kg QW, followed by OP that began after last dose of that treatment cycle. Eligible participants from MG0004 who completed at least 6 scheduled visits for RLZ treatment, PEOT Visit and who were in OP could complete End of Study Visit could move directly into OP in MG0007. These participants underwent their first MG0007 treatment with RLZ upon worsening of MG symptoms. Participants continued their last treatment dose from MG0004. Dose adjustments could be applied in further cycles as per Investigator's discretion. If symptom worsens between assessments, resulting in need for additional treatment, participants underwent another 6-week treatment cycle followed by OP, based on Investigator's discretion.
Period: Overall Study
Arm/Group | Enrolled, But Not Treated | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Started | 8 | 80 | 77
Completed | 3 | 15 | 16
Not Completed | 5 | 65 | 61
Not completed — Adverse Event | 1 | 12 | 14
Not completed — Lack of Efficacy | 1 | 3 | 6
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 17 | 9
Not completed — Last Treatment Per Sponsor Lplv Timelines | 0 | 12 | 6
Not completed — Participant Withdrawn After Drug Approved By FDA | 0 | 0 | 1
Not completed — Pi Withdrew the Patients From the Study | 0 | 0 | 1
Not completed — Withdraw Per Sponsor's Directive | 0 | 1 | 0
Not completed — Withdrawal Due to Prohibited Treatment | 0 | 0 | 1
Not completed — Use of Rescue Medication | 0 | 0 | 1
Not completed — Last Treatment Per Sponsor | 0 | 0 | 2
Not completed — Rescue Medication | 0 | 0 | 1
Not completed — Participant Want to Start a Family | 0 | 0 | 1
Not completed — Withdraw Based on Sponsor Decision | 0 | 0 | 1
Not completed — Participant Screened For MG0020 | 0 | 2 | 3
Not completed — Patient Withdrawn Due To Inappropriate Behavior | 0 | 1 | 0
Not completed — Subject Performed PEOT, Not a Completed Subject | 0 | 1 | 0
Not completed — Participant to Be Screened for MG0020 Study | 0 | 4 | 5
Not completed — End Of Study | 0 | 2 | 1
Not completed — Wish To Continue Study IMP in Patient Programme | 0 | 1 | 0
Not completed — Participant Received Rescue Medication | 0 | 1 | 0
Not completed — Patient Withdrawn; Lack of IMP Shipments | 0 | 2 | 1
Not completed — Last Treatment Per Lplv, Screened For MG0020 | 0 | 2 | 2
Not completed — Discontinued Due to Chronic Heart Failure | 0 | 0 | 1
Not completed — Last Treatment Per Sponsor Lplv Timelines- Japan | 0 | 3 | 3
Not completed — Enrollment Cup | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refers to the Full Analysis set (FAS) which consisted of all enrolled study participants who were randomized in this study or in MG0004.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enrolled, But Not Treated | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg | Total
Number analyzed (Participants) | 8 | 80 | 77 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (17.6) | 52.5 (15.7) | 52.2 (17.0) | 52.7 (16.4)
Age, Customized [Count of Participants; unit: Participants]
  18 to <65 years | 5 | 61 | 57 | 123
  65 to <85 years | 2 | 19 | 19 | 40
  >=85 years | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 45 | 48 | 96
  Male | 5 | 35 | 29 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan native | 0 | 0 | 0 | 0
  Asian | 0 | 8 | 8 | 16
  Black | 3 | 1 | 0 | 4
  Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 1
  White | 4 | 54 | 54 | 112
  Other/mixed | 0 | 0 | 0 | 0
  Missing | 1 | 17 | 14 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 4 | 10
  Not Hispanic or Latino | 3 | 63 | 60 | 126
  Missing | 1 | 15 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which did not necessarily had a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAE was defined as any event that was not present prior to first dose of investigational medicinal product (IMP), or any unresolved event already present that worsened in intensity following treatment, up to 8 weeks after end of Treatment Period or after last dose of IMP in participants who discontinued study or IMP.
Time Frame: From Baseline (Day 1) to End of Study (up to 34 months)
Population: Safety Set (SS): All study participants in the FAS who received at least one dose of IMP. Participants who switched doses were counted in both Rozanolixizumab (RLZ) doses.
Measure: Number; unit: percentage of participants
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 102 | 102
percentage of participants | 78.4 | 94.1

2. Primary Outcome: Percentage of Participants With TEAEs Leading to Withdrawal of Investigational Medicinal Product (IMP)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. AEs leading to permanent withdrawal of study medication.
Time Frame: From Baseline (Day 1) to End of Study (up to 34 months)
Population: Safety Set (SS): All study participants in the FAS who received at least one dose of IMP. Participants who switched doses were counted in both RLZ doses.
Measure: Number; unit: percentage of participants
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 102 | 102
percentage of participants | 9.8 | 16.7

3. Secondary Outcome: Change From Baseline (Day 1) to Day 43 in Myasthenia Gravis-Activities of Daily Living (MG-ADL) Score Within One Treatment Cycle (Cycle 1, 2, and 3)
Description: The MG-ADL is an 8-item PRO instrument developed on basis of QMG. The MG-ADL targeted symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The total MG-ADL score was obtained by summing responses to each individual item (8 items; Grades: 0, 1, 2, 3), where 0= no symptoms or impaired performance and 3= most severe symptoms or impaired performance. The total score ranges from 0 to 24, with higher score indicating more disability. A positive change in score indicates worsening and negative change indicates improvement. For analyses done by study cycle, Baseline values were last available values prior to or on the same date of first administration of IMP at each cycle (Baseline [Day 1]) value for that cycle.
Time Frame: From Baseline (Day 1) to Day 43 of each cycle (Cycles 1, 2, and 3)
Population: Safety Set (SS): All study participants in the FAS who received at least one dose of IMP. Number of Participants Analyzed included those participants who were evaluable for the assessment. Number Analyzed included those participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 74 | 66
score on a scale
  Cycle 1: Treatment (Day 43) | -3.7 (3.5) | -3.1 (2.9)
  Cycle 2: Treatment (Day 43): number analyzed (Participants) | 56 | 65
  Cycle 2: Treatment (Day 43) | -2.9 (3.1) | -3.8 (3.9)
  Cycle 3: Treatment (Day 43): number analyzed (Participants) | 41 | 58
  Cycle 3: Treatment (Day 43) | -3.3 (2.7) | -3.2 (3.3)

4. Secondary Outcome: Change From Baseline (Day 1) to Day 43 in Quantitative Myasthenia Gravis (QMG) Score Within One Treatment Cycle (Cycle 1, 2, and 3)
Description: The QMG is a validated assessment and the scale tested 13 items, including ocular and facial involvement, swallowing, speech, limb strength, and forced vital capacity. The total QMG score was obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3) and the score ranges from 0 to 39, with lower scores indicating lower disease activity. A positive change in the score indicates worsening and a negative change indicates improvement. For the analyses done by study cycle, Baseline values were the last available values prior to or on the same date (and same time if time was collected for the individual assessment) of first administration of IMP at each cycle (ie, Baseline [Day 1]) value for that cycle.
Time Frame: From Baseline (Day 1) to Day 43 of each cycle (Cycles 1, 2, and 3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 73 | 64
score on a scale
  Cycle 1: Treatment (Day 43) | -4.5 (5.0) | -4.1 (4.2)
  Cycle 2: Treatment (Day 43): number analyzed (Participants) | 55 | 64
  Cycle 2: Treatment (Day 43) | -3.9 (4.1) | -4.9 (5.5)
  Cycle 3: Treatment (Day 43): number analyzed (Participants) | 41 | 57
  Cycle 3: Treatment (Day 43) | -5.1 (4.8) | -4.2 (4.4)

5. Secondary Outcome: Change From Baseline (Day 1) to Day 43 in Myasthenia Gravis-Composite (MG-C) Score Within One Treatment Cycle (Cycle 1, 2, and 3)
Description: MG-C scale consists of 10 items which included ptosis (score range=0 to 3), double vision on lateral gaze left/right/both (score range=0 to 4), eye closure (score range=0 to 2), talking (score range=0 to 6), chewing (score range=0 to 6), swallowing (score range=0 to 6), breathing (score range=0 to 9), neck flexion or extension (score range=0 to 4), shoulder abduction (score range=0 to 5) and hip flexion (score range= 0 to 5), lower scores= lower disease activity. Total MG-C score obtained by summing responses to each individual item and score ranges from 0 - 50, (lower scores indicating lower disease activity). Positive change = worsening, and negative change = improvement. For analyses done by study cycle, Baseline values were last available values prior to or on the same date of first administration of IMP at each cycle (Baseline [Day 1]) value for that cycle.
Time Frame: From Baseline (Day 1) to Day 43 of each cycle (Cycles 1, 2, and 3)
Population: Safety Set (SS): All study participants in FAS who received at least 1 dose of IMP. Number of Participants Analyzed included participants who were evaluable for the assessment. Number Analyzed included participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 73 | 66
score on a scale
  Cycle 1: Treatment (Day 43) | -7.6 (7.3) | -4.7 (5.7)
  Cycle 2: Treatment (Day 43): number analyzed (Participants) | 56 | 65
  Cycle 2: Treatment (Day 43) | -5.7 (5.4) | -7.5 (7.0)
  Cycle 3: Treatment (Day 43): number analyzed (Participants) | 41 | 56
  Cycle 3: Treatment (Day 43) | -6.8 (5.9) | -6.1 (7.2)

6. Secondary Outcome: Change From Baseline (Day 1) to Day 43 in Myasthenia Gravis (MG) Symptoms Patient Reported Outcome (PRO) 'Muscle Weakness Fatigability' Score Within One Treatment Cycle (Cycle 1, 2, and 3)
Description: The MG symptoms PRO instrument consisted of 42 items across 5 scales: ocular symptoms (1-5); bulbar muscle weakness (6-15); respiratory muscle weakness (16-18); physical fatigue (19-33) and muscle weakness fatigability (34-42). Study participants had to choose response option that best described severity of ocular, bulbar, and respiratory symptoms over past 7 days using a 4-point Likert scale ("none" to "severe") and frequency of experiencing physical fatigue and muscle weakness fatigability over past 7 days using a 5-point Likert scale (1="none of the time" - 5= "all of the time"), for each item. Sum of each item score is linearly transformed to have all domain scores ranging from 0 to 100, higher scores indicates more severe symptoms. For analyses done by study cycle, Baseline values were last available values prior to or on the same date of first administration of IMP at each cycle (Baseline [Day 1]) value for that cycle.
Time Frame: From Baseline (Day 1) to Day 43 of each cycle (Cycles 1, 2, and 3)
Population: Safety Set (SS): All study participants in FAS who received at least 1 dose of IMP. Number of Participants Analyzed: participants who were evaluable for the assessment. Number Analyzed: participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 75 | 66
score on a scale
  Cycle 1: Treatment (Day 43) | -17.6 (21.0) | -14.6 (17.2)
  Cycle 2: Treatment (Day 43): number analyzed (Participants) | 56 | 65
  Cycle 2: Treatment (Day 43) | -13.2 (19.2) | -19.2 (21.6)
  Cycle 3: Treatment (Day 43): number analyzed (Participants) | 41 | 58
  Cycle 3: Treatment (Day 43) | -12.8 (14.4) | -15.4 (17.7)

7. Secondary Outcome: Change From Baseline (Day 1) to Day 43 in MG Symptoms PRO 'Physical Fatigue' Score Within One Treatment Cycle (Cycle 1, 2, and 3)
Description: The MG symptoms PRO instrument consisted of 42 items across 5 scales: ocular muscle weakness (1-5); bulbar muscle weakness (6-15); respiratory muscle weakness (16-18); physical fatigue (19-33) and muscle weakness fatigability (34-42). Study participants had to choose response option based on frequency of experiencing physical fatigue (19-33) over past 7 days using a 5-point Likert scale (1="none of time" - 5="all of time") for each item. Sum of each item score is linearly transformed to have all domain scores ranging from 0 to 100, higher scores indicated severe symptoms.
Time Frame: From Baseline (Day 1) to Day 43 of each cycle (Cycles 1, 2, and 3)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 75 | 66
score on a scale
  Cycle 1: Treatment (Day 43) | -16.5 (18.6) | -14.8 (18.5)
  Cycle 2: Treatment (Day 43): number analyzed (Participants) | 56 | 65
  Cycle 2: Treatment (Day 43) | -13.6 (21.6) | -16.0 (18.2)
  Cycle 3: Treatment (Day 43): number analyzed (Participants) | 41 | 58
  Cycle 3: Treatment (Day 43) | -15.3 (16.9) | -15.0 (18.4)

8. Secondary Outcome: Change From Baseline (Day 1) to Day 43 in MG Symptoms PRO 'Bulbar Muscle Weakness' Score Within One Treatment Cycle (Cycle 1, 2, and 3)
Description: The MG symptoms PRO instrument consisted of 42 items across 5 scales: ocular muscle weakness (1-5); bulbar muscle weakness (6-15); respiratory muscle weakness (16-18); physical fatigue (19-33) and muscle weakness fatigability (34-42). Bulbar symptoms are now recognised as bulbar muscle weakness. Study participants were asked to choose response option that best described severity of bulbar muscle weakness (6-15) symptoms over past 7 days using a 4-point Likert scale (1="none" to 4="severe") for each item. Sum of each item score is linearly transformed to have all domain scores ranging from 0 to 100, higher scores indicated severe symptoms.
Time Frame: From Baseline (Day 1) to Day 43 of each cycle (Cycles 1, 2, and 3)
Population: Safety Set (SS): All study participants in the FAS who received at least one dose of IMP. Number of Participants Analyzed: participants who were evaluable for the assessment. Number Analyzed included those participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 75 | 66
score on a scale
  Cycle 1: Treatment (Day 43) | -13.4 (19.8) | -11.6 (16.2)
  Cycle 2: Treatment (Day 43): number analyzed (Participants) | 56 | 65
  Cycle 2: Treatment (Day 43) | -10.4 (16.2) | -15.5 (18.1)
  Cycle 3: Treatment (Day 43): number analyzed (Participants) | 41 | 58
  Cycle 3: Treatment (Day 43) | -14.0 (16.8) | -13.0 (17.9)

9. Secondary Outcome: MG-ADL Responder Rate (>=2.0-point Improvement From Baseline [Day 1]) Within One Treatment Cycle (Cycle 1, 2, and 3 [Day 43])
Description: The MG-ADL is an 8-item PRO instrument developed on the basis of the Quantitative Myasthenia Gravis (QMG). The MG-ADL targeted symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The total MG-ADL score was obtained by summing the responses to each individual item (8 items; Grades: 0, 1, 2, 3), where 0 represents no symptoms or impaired performance and 3 represents the most severe symptoms or impaired performance. The total score ranges from 0 to 24, with a higher score indicating more disability. A MG-ADL responder was defined as achieving at least 2.0-point improvement (decrease) in the MG-ADL score from Baseline.
Time Frame: Day 43 of Cycle 1, 2, and 3
Population: Safety Set (SS): All study participants in the FAS who received at least one dose of IMP. Number of Participants Analyzed included those participants who were evaluable for the assessment. Number Analyzed: participants who were evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 74 | 66
percentage of participants
  Cycle 1: Treatment (Day 43) | 74.3 | 63.6
  Cycle 2: Treatment (Day 43): number analyzed (Participants) | 56 | 65
  Cycle 2: Treatment (Day 43) | 62.5 | 67.7
  Cycle 3: Treatment (Day 43): number analyzed (Participants) | 41 | 58
  Cycle 3: Treatment (Day 43) | 73.2 | 67.2

10. Secondary Outcome: Time to MG-ADL Response (>=2.0-point Improvement From Baseline [Day 1]) Within One Treatment Cycle (Cycle 1, 2, and 3)
Description: Time to achieve MG-ADL response, defined as at least 2.0-point improvement from Baseline. Time to first MG-ADL response (in days) by study cycle was defined as date of first MG-ADL Response within study cycle - date of MG-ADL Baseline within study cycle + 1.
Time Frame: From Baseline (Day 1) to Day 43 of each cycle (Cycles 1, 2, and 3)
Population: Safety Set (SS): All study participants in the FAS who received at least one dose of IMP. Number Analyzed: participants who were evaluable at specified timepoint.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 80 | 77
days
  Cycle 1 | 9.00 [8.00 to 15.00] | 22.00 [15.00 to 36.00]
  Cycle 2: number analyzed (Participants) | 59 | 67
  Cycle 2 | 15.00 [10.00 to 17.00] | 15.00 [9.00 to 22.00]
  Cycle 3: number analyzed (Participants) | 44 | 61
  Cycle 3 | 15.00 [9.00 to 15.00] | 15.00 [9.00 to 17.00]

11. Secondary Outcome: Time Between Consecutive Treatment Cycles
Description: Time between consecutive treatment cycles: Study participants were assessed for MG worsening prior to repeated cycles. In case of symptom worsening (eg, an increase of 2.0 points on MG-ADL or 3.0 points on QMG scale) between assessments, resulted additional treatment, study participants undergone another 6-week treatment cycle followed by an Observation Period, based on Investigator's discretion. Time between treatment cycles was calculated as: date of first sc infusion in consecutive cycle - date of last sc infusion before new cycle + 1 (or date of censoring - date of last sc infusion before potential new cycle + 1).
Time Frame: From end of the 6-week treatment cycle (Day 43) to the next 6-week treatment cycle (Day 1), assessed up to 2.5 years
Population: Safety Set (SS): All study participants in FAS who received at least 1 dose of IMP. Number Analyzed: participants who were evaluable at specified timepoint.
Measure: Median (Full Range); unit: days
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 80 | 77
days
  Between Cycle 1 and Cycle 2 | 64.0 [9 to 883] | 51.0 [2 to 856]
  Between Cycle 2 and Cycle 3: number analyzed (Participants) | 59 | 67
  Between Cycle 2 and Cycle 3 | 58.0 [1 to 631] | 50.0 [15 to 575]
  Between Cycle 3 and Cycle 4: number analyzed (Participants) | 44 | 61
  Between Cycle 3 and Cycle 4 | 42.5 [27 to 399] | 43.0 [5 to 194]
  Between Cycle 4 and Cycle 5: number analyzed (Participants) | 40 | 55
  Between Cycle 4 and Cycle 5 | 43.0 [9 to 181] | 43.0 [17 to 242]
  Between Cycle 5 and Cycle 6: number analyzed (Participants) | 36 | 51
  Between Cycle 5 and Cycle 6 | 44.0 [22 to 192] | 43.0 [15 to 175]
  Between Cycle 6 and Cycle 7: number analyzed (Participants) | 33 | 49
  Between Cycle 6 and Cycle 7 | 36.0 [8 to 348] | 43.0 [7 to 106]
  Between Cycle 7 and Cycle 8: number analyzed (Participants) | 31 | 40
  Between Cycle 7 and Cycle 8 | 37.0 [22 to 87] | 37.0 [6 to 84]
  Between Cycle 8 and Cycle 9: number analyzed (Participants) | 27 | 36
  Between Cycle 8 and Cycle 9 | 36.0 [8 to 120] | 36.0 [7.0 to 134]
  Between Cycle 9 and Cycle 10: number analyzed (Participants) | 21 | 31
  Between Cycle 9 and Cycle 10 | 29.0 [7 to 97] | 29.0 [8 to 72]
  Between Cycle 10 and Cycle 11: number analyzed (Participants) | 15 | 26
  Between Cycle 10 and Cycle 11 | 29.0 [8 to 64] | 29.0 [8 to 99]
  Between Cycle 11 and Cycle 12: number analyzed (Participants) | 11 | 19
  Between Cycle 11 and Cycle 12 | 23.0 [8 to 52] | 22.0 [7 to 37]
  Between Cycle 12 and Cycle 13: number analyzed (Participants) | 9 | 13
  Between Cycle 12 and Cycle 13 | 22.0 [6 to 36] | 22.0 [7 to 38]
  Between Cycle 13 and Cycle 14: number analyzed (Participants) | 5 | 9
  Between Cycle 13 and Cycle 14 | 29.0 [22 to 35] | 16.0 [8 to 65]
  Between Cycle 14 and Cycle 15: number analyzed (Participants) | 4 | 5
  Between Cycle 14 and Cycle 15 | 29.0 [29 to 64] | 9.0 [8 to 16]
  Between Cycle 15 and Cycle 16: number analyzed (Participants) | 3 | 2
  Between Cycle 15 and Cycle 16 | 23.0 [8 to 29] | 26.5 [9 to 44]
  Between Cycle 16 and Cycle 17: number analyzed (Participants) | 1 | 0
  Between Cycle 16 and Cycle 17 | 29.0 [29 to 29] |
  Between Cycle 17 and Cycle 18: number analyzed (Participants) | 1 | 0
  Between Cycle 17 and Cycle 18 | 8.0 [8 to 8] |

ADVERSE EVENTS:
Time Frame: Enrolled, but not treated: From Screening until End of Study (up to 34 months); Randomized participants: From Baseline (Day 1) until End of Study (up to 34 months)
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with use of study medication, whether or not considered related to study medication. TEAEs were reported for all study participants in the FAS who received at least 1 dose of IMP. Eligible participants who did not undergo any treatment of RLZ but experienced an AE, are presented in a separate group "Enrolled but not treated". Participants who switched doses were counted in both RLZ doses.
Arm/Group | Enrolled, But Not Treated | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/8 | 1/102 | 3/102
Serious Adverse Events (participants affected / at risk) | 3/8 | 16/102 | 31/102
Other Adverse Events (participants affected / at risk) | 5/8 | 67/102 | 78/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled, But Not Treated (N=8) | Rozanolixizumab ~7 mg/kg (N=102) | Rozanolixizumab ~10 mg/kg (N=102)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal disorder (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis aspergillus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 5 (8) | 11 (17)
Myasthenia gravis crisis (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Subacute cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thymectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled, But Not Treated (N=8) | Rozanolixizumab ~7 mg/kg (N=102) | Rozanolixizumab ~10 mg/kg (N=102)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 20 (49) | 28 (55)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 10 (11) | 7 (11)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 6 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 9 (17) | 18 (26)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 8 (10)
COVID-19 (Infections and infestations) | 1 (1) | 15 (15) | 24 (26)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 7 (13) | 11 (22)
Nasopharyngitis (Infections and infestations) | 1 (1) | 10 (16) | 11 (14)
Urinary tract infection (Infections and infestations) | 1 (1) | 6 (12) | 2 (3)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 7 (10)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 8 (9)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 6 (13) | 15 (27)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 6 (10)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (8) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 12 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 6 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (7) | 8 (8)
Headache (Nervous system disorders) | 0 (0) | 36 (99) | 46 (218)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 10 (11)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 2 (2) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 6 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 9 (13)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 8 (11)
Pyrexia (General disorders) | 0 (0) | 9 (20) | 19 (34)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 7 (8)
Oedema peripheral (General disorders) | 0 (0) | 7 (8) | 8 (9)
Hepatic pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 5 (6)
Interferon gamma release assay positive (Investigations) | 1 (1) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT04650854/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT04650854/SAP_001.pdf